CLINICAL TRIAL: NCT07396051
Title: A Randomized Controlled Trial of Multimodal Rehabilitation Versus Standard Care on Adjacent Segment Degeneration in Frail Elderly Patients Undergoing Short-Segment Lumbar Fusion
Brief Title: Rehabilitation Exercise Against Complications in High-risk Elderly After Lumbar Fusion(REACH)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Xuanwu-REACH
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Adjacent Segment Degeneration; Multimodal Rehabilitation; Lumber Fusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Care Group (No Intervention): All patients in this group undergo standard Enhanced Recovery After Surgery (ERAS) protocols tailored for frail individuals, which encompass optimization of nutrition, pain management, early mobilization, and other evidence-based perioperative measures.
- Multimodal Rehabilitation Group (Experimental): This group receives a supervised, structured, and progressive multimodal rehabilitation program in addition to the standard perioperative Enhanced Recovery After Surgery (ERAS) care and initial home exercise guidance.
  Interventions: Behavioral: Postoperative Multimodal Rehabilitation Program

INTERVENTIONS:
Behavioral: Postoperative Multimodal Rehabilitation Program — All subjects independently completed the training program postoperatively. During follow-up, two physical therapists were responsible for arranging and designing the training sessions for the next phase. The therapists possessed equivalent levels of clinical experience. Based on clinical experience, scientific knowledge, and personal conviction, the therapists were confident that they provided the best treatment plan for the patients. To ensure consistency in treatment implementation throughout the study, fidelity checks were conducted at the end of each treatment session and course, in accordance with the cognitive-behavioral therapy and exercise training implementation manual. After enrollment, patients did not receive other treatments (such as physical therapy or nerve block), and the use of major pharmacological agents was prohibited, except for the allowance of mild analgesics and non-steroidal anti-inflammatory drugs.
  Arms: Multimodal Rehabilitation Group

SUMMARY:
This is a prospective, randomized controlled trial aimed at evaluating whether a structured multimodal rehabilitation program can delay or reduce the occurrence of adjacent segment degeneration (ASDeg) in frail elderly patients after short-segment lumbar fusion surgery.

DETAILED DESCRIPTION:
Background and Rationale Adjacent segment degeneration (ASDeg) is a well-recognized long-term complication following lumbar fusion surgery. Frail elderly patients, characterized by diminished physiological reserve and increased vulnerability to stressors, represent a growing surgical population with a potentially higher risk for poor postoperative outcomes, including accelerated ASDeg. While enhanced recovery after surgery (ERAS) protocols have improved short-term recovery, there is a significant lack of evidence regarding structured, long-term rehabilitation strategies aimed at modifying the disease progression and functional decline in this high-risk group postoperatively. This study hypothesizes that a supervised, multimodal rehabilitation program initiated after the initial postoperative healing phase will improve spinal stability, muscle function, and overall physical resilience, thereby delaying the onset of ASDeg and improving functional outcomes compared to standard care alone.

Study Objectives Primary Objective: To compare the time to the development of radiographically confirmed adjacent segment degeneration between frail elderly patients receiving a multimodal rehabilitation program and those receiving standard care after short-segment lumbar fusion.

Secondary Objectives: To compare the two groups regarding: The incidence of ASDeg at 2 years postoperatively.

Changes in patient-reported outcomes: back and leg pain Visual Analog Scale (VAS), Oswestry Disability Index (ODI), and lumbar Japanese Orthopaedic Association (JOA) score. Changes in frailty status (Fried score) and bone mineral density (BMD). Radiographic parameters including sagittal vertical axis (SVA), pelvic incidence-lumbar lordosis mismatch (PI-LL), and segmental angles.

Study Design This is a prospective, randomized, controlled, parallel-group, superiority trial with an assessor-blinded outcome evaluation.

Participants

Inclusion Criteria:

Age ≥ 75 years. Classified as "frail" according to the Fried frailty phenotype. Scheduled for first-time, posterior short-segment (1-2 levels) lumbar instrumented fusion surgery. Willing and able to provide written informed consent and complete the 2-year follow-up.

Exclusion Criteria:

History of previous lumbar spine surgery. Lumbar pathology due to tumor, trauma, infection, or congenital deformity. Comorbidities with a severe impact on prognosis or ability to participate in rehabilitation (e.g., severe cardiopulmonary disease, advanced dementia).

Interventions All Participants: Receive standard perioperative ERAS management. Prior to discharge, all patients receive a single 30-minute instruction session for a home-based program encouraging walking, and light abdominal, back, and thigh muscle strengthening, along with hip stretching.

Control Group (Standard Care): Receive no further structured intervention beyond the initial home program guidance and routine clinical follow-up.

Intervention Group (Multimodal Rehabilitation): In addition to standard care, participants commence a supervised, progressive rehabilitation program at 12 weeks postoperatively. The program lasts 48 weeks and consists of:

Weekly remote adherence monitoring via phone or a dedicated app using a Likert scale (1-4 points per week).

Periodic in-person clinical visits with a physiotherapist for exercise progression, technique correction, and provision of illustrated training manuals for the next phase.

Good adherence is defined as a cumulative score >135 points (out of a maximum 196, >70%).

Outcome Measures Primary Outcome: Time (in days) from surgery to the development of adjacent segment degeneration on imaging. Data for patients without ASDeg will be censored at 730 days (2 years).

Secondary Outcomes: Assessed at preoperative, postoperative immediate, 12, 24, 48, 60, 72, and 96 weeks.

Incidence of ASDeg at 2 years. VAS (back/leg), ODI, JOA scores, Fried Frailty Score, Bone Mineral Density (BMD). Radiographic parameters: Disc height, Cobb angle, Modic changes, SVA, PI, PT, SS, LL, PI-LL.

Sample Size Calculation The sample size was calculated using G*Power 3.1.9.7 software. Assuming a Cohen's d effect size of 0.5, a two-sided alpha of 0.05, and a power of 0.95 (1-β) for an independent t-test, 88 participants per group are required. Accounting for an estimated 20% dropout/loss to follow-up rate, the final sample size is 106 participants per group, for a total of 212 participants.

Statistical Analysis Primary Analysis: The primary outcome will be analyzed using Kaplan-Meier survival curves and compared between groups using the log-rank test. A Cox proportional hazards model will be used to calculate hazard ratios.

General Principles: Analyses will follow the Intent-to-Treat (ITT) principle. Missing data will be handled using the Last Observation Carried Forward (LOCF) method.

Secondary Analyses: Continuous variables will be compared using independent t-tests or Mann-Whitney U tests based on normality (assessed by Kolmogorov-Smirnov test). Categorical variables will be compared using Chi-square or Fisher's exact test. Data will be presented as mean (SD), median (IQR), or n (%).

Sensitivity/Exploratory Analyses: Sensitivity analyses (e.g., per-protocol) and exploratory mediator analyses are planned to assess robustness and potential mechanisms.

Data Collection and Management Data will be collected prospectively using standardized case report forms (CRFs), including demographics, clinical scores, and radiographic measurements. All data will be stored in a secure, password-protected database.

Ethics and Dissemination The study protocol will be submitted for approval to the relevant Institutional Review Board / Ethics Committee prior to initiation. Written informed consent will be obtained from all participants. The results of this trial will be disseminated through peer-reviewed publications and conference presentations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 years.
* Classified as "frail" according to the Fried frailty phenotype.
* Scheduled for first-time, posterior short-segment (1-2 levels) lumbar instrumented fusion surgery.
* Willing and able to provide written informed consent and complete the 2-year follow-up.

Exclusion Criteria:

* History of previous lumbar spine surgery.
* Lumbar pathology due to tumor, trauma, infection, or congenital deformity.
* Comorbidities with a severe impact on prognosis or ability to participate in rehabilitation (e.g., severe cardiopulmonary disease, advanced dementia).

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Time to Adjacent Segment Degeneration (ASDeg) | From surgery date up to 2 years postoperatively (730 days).
  The number of days from the surgery date to the radiographic diagnosis of ASDeg. For participants who do not develop ASD during the study, the data will be censored at 730 days (2 years postoperatively). This measure is used to compare the intervention and control groups.

SECONDARY OUTCOMES:
Comprehensive Complication Index | Preoperative; immediately postoperative; and at 12, 24, 48, 60, 72, and 96 weeks postoperatively.
  The Comprehensive Complication Index (CCI) is based on the complication grading by the Clavien-Dindo Classification and captures every complication that occurred after an intervention. Postoperative complications were recorded to 90-day after surgery (definitions provided in supplementary table 1) and scored by severity using the Clavien-Dindo classification. The CCI was derived from these scores using the CCI calculator available online (http://www.assessurgery.com). Previous studies have validated the CCI as a measure of postoperative morbidity, suggesting that it offers a more comprehensive and sensitive endpoint for surgical research compared to traditional morbidity measures, such as the overall rate of complications or the rate of severe complications.
Oswestry disability index | Preoperative; immediately postoperative; and at 12, 24, 48, 60, 72, and 96 weeks postoperatively.
  Oswestry disability index (0 - 100 points, a higher total score reflects higher disability) for lumbar surgery.
Leg Pain Visual Analog Scale (VAS) Score | Preoperative; immediately postoperative; and at 12, 24, 48, 60, 72, and 96 weeks postoperatively.
  Patient-reported intensity of leg pain (radicular pain) measured on Visual Analog Scale (VAS), where 0 represents "no pain" and 10 represents "worst imaginable pain".
Japanese Orthopaedic Association (JOA) Score for Low Back Pain | Preoperative; immediately postoperative; and at 12, 24, 48, 60, 72, and 96 weeks postoperatively.
  Clinician-assessed lumbar spine function measured by the Japanese Orthopaedic Association (JOA) score. Higher scores indicate better function.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing 10034, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gillis C, Ljungqvist O, Carli F. Prehabilitation, enhanced recovery after surgery, or both? A narrative review. Br J Anaesth. 2022 Mar;128(3):434-448. doi: 10.1016/j.bja.2021.12.007. Epub 2022 Jan 7. PMID 35012741
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Parker SG, McCue P, Phelps K, McCleod A, Arora S, Nockels K, Kennedy S, Roberts H, Conroy S. What is Comprehensive Geriatric Assessment (CGA)? An umbrella review. Age Ageing. 2018 Jan 1;47(1):149-155. doi: 10.1093/ageing/afx166. PMID 29206906
- [Background] Whittle AK, Kalsi T, Babic-Illman G, Wang Y, Fields P, Ross PJ, Maisey NR, Hughes S, Kwan W, Harari D. A comprehensive geriatric assessment screening questionnaire (CGA-GOLD) for older people undergoing treatment for cancer. Eur J Cancer Care (Engl). 2017 Sep;26(5). doi: 10.1111/ecc.12509. Epub 2016 May 1. PMID 27132979
- [Background] Karsy M, Chan AK, Mummaneni PV, Virk MS, Bydon M, Glassman SD, Foley KT, Potts EA, Shaffrey CI, Shaffrey ME, Coric D, Asher AL, Knightly JJ, Park P, Fu KM, Slotkin JR, Haid RW, Wang M, Bisson EF. Outcomes and Complications With Age in Spondylolisthesis: An Evaluation of the Elderly From the Quality Outcomes Database. Spine (Phila Pa 1976). 2020 Jul 15;45(14):1000-1008. doi: 10.1097/BRS.0000000000003441. PMID 32097272
- [Background] Martin BI, Mirza SK, Spina N, Spiker WR, Lawrence B, Brodke DS. Trends in Lumbar Fusion Procedure Rates and Associated Hospital Costs for Degenerative Spinal Diseases in the United States, 2004 to 2015. Spine (Phila Pa 1976). 2019 Mar 1;44(5):369-376. doi: 10.1097/BRS.0000000000002822. PMID 30074971
- [Background] Rivier C, Shen GH. In the rat, endogenous nitric oxide modulates the response of the hypothalamic-pituitary-adrenal axis to interleukin-1 beta, vasopressin, and oxytocin. J Neurosci. 1994 Apr;14(4):1985-93. doi: 10.1523/JNEUROSCI.14-04-01985.1994. PMID 8158253
- [Background] Kassebaum DG, Judkins MP, Griswold HE. Stress electrocardiography in the evaluation of surgical revascularization of the heart. Circulation. 1969 Sep;40(3):297-313. doi: 10.1161/01.cir.40.3.297. No abstract available. PMID 5810888